CLINICAL TRIAL: NCT02357147
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of Amatuximab in Combination With Pemetrexed and Cisplatin in Subjects With Unresectable Malignant Pleural Mesothelioma
Brief Title: Study of the Safety and Efficacy of Amatuximab in Combination With Pemetrexed and Cisplatin in Subjects With Unresectable Malignant Pleural Mesothelioma (MPM)
Acronym: ARTEMIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to business reasons
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MORAb-009-201; 2014-004489-85 (EudraCT Number)
Record Dates: First submitted 2015-01-14; First posted 2015-02-06 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2017-02

CONDITIONS: Mesothelioma, Malignant
Keywords: Amatuximab; Pemetrexed; Cisplatin; Unresectable Malignant Pleural Mesothelioma; ARTEMIS
MeSH Terms: conditions — Mesothelioma, Malignant; Severe combined immunodeficiency with sensitivity to ionizing radiation | interventions — amatuximab; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Combination Phase - Amatuximab + Pemetrexed and Cisplatin
  Maintenance Phase - Amatuximab
  Interventions: Drug: Amatuximab; Drug: Pemetrexed; Drug: Cisplatin
- Arm 2 (Experimental): Combination Phase - Placebo + Pemetrexed and Cisplatin
  Maintenance Phase - Placebo
  Interventions: Drug: Placebo; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Placebo — Combination Phase - Placebo will be administered IV (intravenous infusion) once weekly for six 21-day cycles.
  Maintenance Phase - Placebo will be administered IV (intravenous infusion) once weekly until disease progression.
  Arms: Arm 2
Drug: Amatuximab — Combination Phase - Amatuximab 5mg/kg will be administered IV (intravenous infusion) once weekly for six 21-day cycles.
  Maintenance Phase - Amatuximab 5mg/kg will be administered IV (intravenous infusion) once weekly until disease progression.
  Arms: Arm 1
Drug: Pemetrexed — Combination Phase - Pemetrexed 500 mg/m^2 will be administered IV on Day 1 of each 21-day cycle for 6 cycles.
Drug: Cisplatin — Combination Phase - Cisplatin 75 mg/m^2 will be administered IV on Day 1 of each 21-day cycle for 6 cycles.

SUMMARY:
This study was originally designed as a multicenter, double-blind, randomized, parallel-group study, using a placebo control or amatuximab 5 milligrams per kilogram (mg/kg), administered weekly, designed to evaluate the safety and efficacy of amatuximab in combination with pemetrexed and cisplatin in participants with unresectable Malignant Pleural Mesothelioma (MPM) who have not received prior systemic therapy.

Per a business decision made by the Sponsor, participants who were randomized to amatuximab and were still on active treatment at the time of the protocol amendment may have consented to continue to receive weekly treatment with amatuximab until disease progression or intolerable toxicity at the discretion of the principal investigator. Participants randomized to placebo or who were in follow-up at the time of the amendment have been discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age at the time of informed consent
2. Have confirmed diagnosis of MPM with the following characteristics:

   * Unresectable disease (defined as the participant not being a candidate for curative surgery)
   * Epithelial type
   * Have an archived tissue sample to be submitted either as a formalin fixed paraffin-embedded (FFPE) tumor block, or 5 to 15 unstained slides
3. Have measurable disease at Screening by computed tomography (CT) (or magnetic resonance imaging [MRI]) as defined by at least 1 lesion of greater than or equal to 1.5 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to the modified RECIST criteria
4. Have other significant medical conditions well-controlled and stable in the opinion of the investigator for at least 30 days prior to Day 1
5. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1 at Screening
6. Have a life expectancy of at least 3 months, as estimated by the investigator
7. Have adequate organ reserve as determined by laboratory test results obtained within 2 weeks prior to Study Day 1 as indicated below:

   * Absolute neutrophil count greater than or equal to 1.5 x 10^9/L
   * Platelet count greater than or equal to 100 x 10^9/L
   * Hemoglobin greater than or equal to 9 g/dL
   * Serum bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (Participants with serum bilirubin abnormalities greater than this specified limit are eligible only if they have known Gilberts disease)
   * Aspartate aminotransferase less than or equal to 3 x ULN
   * Alanine aminotransferase less than or equal to 3 x ULN
   * Alkaline phosphatase less than or equal to 3 x ULN
8. Have a calculated serum creatinine clearance greater than or equal to 45 mL/min using the Cockcroft-Gault equation
9. Participants of childbearing potential must be surgically sterile or consent to use a highly effective method of contraception throughout the study period. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). If a participant of childbearing potential is neither surgically sterile nor postmenopausal, highly effective contraceptive measures must start either prior to or at Screening and continue throughout the entire study period and for at least 6 months after the last dose of chemotherapy and at least 30 days after the last dose of Test Article (amatuximab or placebo) is administered (whichever is later). A highly effective method of contraception is defined as one that results in a low failure rate (that is, less than 1% per year) when used consistently and correctly. Periodic abstinence, the rhythm method, the withdrawal method, condoms, and diaphragms are not acceptable methods of contraception. Women of childbearing potential must also refrain from egg cell donation for 6 months after the final dose of investigational product
10. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period and for 6 months after discontinuation of chemotherapy and for 5 weeks after Test Article (amatuximab or placebo) discontinuation (whichever is later). No sperm donation is allowed during the study period and for 90 days after Test Article discontinuation
11. Be willing and able to provide written informed consent
12. Be willing and able to comply with all aspects of the protocol
13. Participants who were enrolled in the study and randomized to the amatuximab treatment arm may, at the discretion of the principle investigator (PI), consent to continue to receive amatuximab therapy until disease progression, intolerable toxicity, or withdraw of consent

Exclusion Criteria:

1. Have any history of the following:

   * Prior systemic therapy or radiotherapy for MPM; local radiotherapy of noncurative intent (ie, for prevention of instrument-tract recurrence and/or symptom control) is permitted
   * Evidence of other active, invasive malignancy requiring treatment within the past 5 years; noninvasive cancer history (such as carcinoma-in-situ [CIS] that has been resected) is allowed
2. Currently have mesothelioma of the sarcomatous type, mixed histologic disease, or have malignant peritoneal mesothelioma
3. Have confirmed presence of central nervous system metastases
4. Active viral hepatitis or active human immunodeficiency virus infection
5. Have evidence of any other serious systemic disease, including active bacterial or fungal infection, or any medical condition that, in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
6. Clinically significant heart disease (eg, congestive heart failure of New York Heart Association Class 3 or 4, angina not well controlled by medication, or myocardial infarction within 6 months)
7. Electrocardiogram (ECG) demonstrating clinically significant arrhythmias (Note: participants with chronic atrial arrhythmia, ie, atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible). A clinically significant ECG abnormality, including a marked prolonged QT/QTc interval (eg, a repeated demonstration of a QTc interval of greater than 500 ms)
8. Have known intolerance to the Test Article (ie, documented hypersensitivity AE to prior monoclonal antibody therapy, or to amatuximab or any of its excipients)
9. Pregnant and/or lactating females are excluded; a negative beta-human chorionic gonadotropin [B-hCG]) is required during Screening, and a separate local assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of Test Article
10. Have any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study
11. Are scheduled for debulking surgery during the study
12. Are currently enrolled in another clinical study or used any investigational drug or device within 30 days (or 5 x the half-life of the investigational drug/device, whichever is longer) preceding informed consent
13. Participants previously randomized to placebo
14. Participants who have not signed the updated informed consent form associated with this amendment 2
15. Participants who have radiographic or clinical disease progression or intolerable toxicity such that ongoing amatuximab treatment through this study is not appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (7):
  - La Jolla, California
  - Newark, Delaware
  - Bethesda, Maryland
  - Rochester, Minnesota
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Spokane, Washington
- Australia (4):
  - Camperdown, New South Wales
  - Auchenflower, Queensland
  - Richmond, Victoria
  - Perth, Western Australia
- France (8):
  - Caen
  - Créteil
  - La Tronche
  - Lille
  - Lyon
  - Marseille
  - Rennes
  - Toulouse
- Germany (9):
  - Berlin
  - Esslingen am Neckar
  - Frankfurt am Main
  - Gauting
  - Hamburg
  - Hanover
  - Löwenstein
  - Ulm
  - Wöhrendamm
- Italy (11):
  - Rozzano, Milano
  - Pisa, Paradisa 2
  - Alessandria
  - Aviano
  - Bari
  - Bergamo
  - Genoa
  - Genova
  - Monza
  - Orbassano
  - Parma
- United Kingdom (10):
  - Maidstone, Kent
  - Dundee
  - Hereford
  - Leicester
  - London
  - Middlesex
  - Preston
  - Southampton
  - Swindon
  - Taunton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 36 investigative sites in the United States, France, Germany, Italy, the United Kingdom, and Australia from 03 November 2015 to 30 November 2018.
Pre-assignment Details: A total of 124 participants were enrolled (signed informed consent form), of which, 16 were screen failures, 108 were randomized, and 106 were treated. Deaths that were primary cause of treatment discontinuation are reported in participant flow excluding those that occurred after treatment discontinuation.
Groups:
- Amatuximab + Pemetrexed + Cisplatin: During Combination Treatment Phase, participants received amatuximab 5 milligram per kilogram (mg/kg), infusion, intravenously, once weekly in 21-day cycles and pemetrexed 500 milligram per square meter (mg/m^2) and cisplatin 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-day cycle for 6 cycles. Following completion of the Combination Treatment Phase, participants who had not progressed entered the Maintenance Phase and continued to receive amatuximab 5 mg/kg, infusion, intravenously, once weekly until disease progression.
- Placebo + Pemetrexed + Cisplatin: During Combination Treatment Phase, participants received placebo matched to amatuximab infusion, intravenously, once weekly in 21-day cycles and pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-day cycle for 6 cycles. Following completion of the Combination Treatment Phase, participants who had not progressed entered the Maintenance Phase and received placebo matched to amatuximab infusion, intravenously, once weekly until disease progression.
Period: Combination Treatment Phase
Arm/Group | Amatuximab + Pemetrexed + Cisplatin | Placebo + Pemetrexed + Cisplatin
Started | 52 | 56
Treated | 52 | 54
Completed | 26 | 29
Not Completed | 26 | 27
Not completed — Progressive Disease (Radiographic test) | 3 | 3
Not completed — Progressive Disease(Clinical assessment) | 0 | 1
Not completed — Investigator Discretion | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Test Article Held (Greater than 21 Days) | 4 | 1
Not completed — Adverse Event | 12 | 4
Not completed — Death | 1 | 1
Not completed — Sponsor Decision | 0 | 12
Not completed — Other | 1 | 0
Not completed — Not treated | 0 | 2
Period: Maintenance Treatment Phase
Arm/Group | Amatuximab + Pemetrexed + Cisplatin | Placebo + Pemetrexed + Cisplatin
Started | 26 | 29
Treated | 25 | 29
Completed | 0 | 0
Not Completed | 26 | 29
Not completed — Progressive Disease (Radiographic test) | 15 | 10
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Test Article Held (Greater than 21 Days) | 10 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Sponsor Decision | 0 | 15
Not completed — Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all randomized participants who received at least 1 dose of study drug.
Groups:
- Amatuximab + Pemetrexed + Cisplatin: During Combination Treatment Phase, participants received amatuximab 5 mg/kg, infusion, intravenously, once weekly in 21-day cycles and pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-day cycle for 6 cycles. Following completion of the Combination Treatment Phase, participants who had not progressed entered the Maintenance Phase and continued to receive amatuximab 5 mg/kg, infusion, intravenously, once weekly until disease progression.
- Total: Total of all reporting groups
Arm/Group | Amatuximab + Pemetrexed + Cisplatin | Placebo + Pemetrexed + Cisplatin | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (6.08) | 66.9 (7.96) | 67.4 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 37 | 40 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 42 | 37 | 79
  Unknown or Not Reported | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 45 | 46 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs included both non-SAEs and SAEs and the same participant can have both SAEs and as well non-SAEs.
Time Frame: Baseline up to 3 years
Population: The safety analysis set was defined as all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Combination Treatment Phase:Amatuximab + Pemetrexed +Cisplatin: During Combination Treatment Phase, participants received amatuximab 5 mg/kg, infusion, intravenously, once weekly in 21-day cycles and pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-day cycle for 6 cycles.
- Combination Treatment Phase: Placebo + Pemetrexed + Cisplatin: During Combination Treatment Phase, participants received placebo matched to amatuximab infusion, intravenously, once weekly in 21-day cycles and pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-day cycle for 6 cycles.
- Maintenance Treatment Phase: Amatuximab: Following completion of the Combination Treatment Phase, participants who had not progressed entered the Maintenance Phase and continued to receive amatuximab 5 mg/kg, infusion, intravenously, once weekly until disease progression.
- Maintenance Treatment Phase: Placebo: Following completion of the Combination Treatment Phase, participants who had not progressed entered the Maintenance Phase and received placebo matched to amatuximab infusion, intravenously, once weekly until disease progression.
Arm/Group | Combination Treatment Phase:Amatuximab + Pemetrexed +Cisplatin | Combination Treatment Phase: Placebo + Pemetrexed + Cisplatin | Maintenance Treatment Phase: Amatuximab | Maintenance Treatment Phase: Placebo
Number analyzed (Participants) | 52 | 54 | 25 | 29
Participants
  AEs | 50 | 52 | 19 | 21
  SAEs | 15 | 11 | 1 | 4

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug or until date of death (approximately up to 3 years)
Description: Deaths that happened anytime during the study (including those during the treatment and after treatment discontinuation) are reported in this section.
Arm/Group | Combination Treatment Phase:Amatuximab + Pemetrexed +Cisplatin | Combination Treatment Phase: Placebo + Pemetrexed + Cisplatin | Maintenance Treatment Phase: Amatuximab | Maintenance Treatment Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 6/52 | 3/54 | 2/25 | 1/29
Serious Adverse Events (participants affected / at risk) | 15/52 | 11/54 | 1/25 | 4/29
Other Adverse Events (participants affected / at risk) | 50/52 | 51/54 | 19/25 | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Treatment Phase:Amatuximab + Pemetrexed +Cisplatin (N=52) | Combination Treatment Phase: Placebo + Pemetrexed + Cisplatin (N=54) | Maintenance Treatment Phase: Amatuximab (N=25) | Maintenance Treatment Phase: Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amaurosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Treatment Phase:Amatuximab + Pemetrexed +Cisplatin (N=52) | Combination Treatment Phase: Placebo + Pemetrexed + Cisplatin (N=54) | Maintenance Treatment Phase: Amatuximab (N=25) | Maintenance Treatment Phase: Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 11 (29) | 12 (21) | 3 (11) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 13 (35) | 10 (28) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (6) | 3 (4) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (5) | 5 (5) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (27) | 22 (32) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 11 (17) | 10 (13) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 9 (10) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (78) | 39 (83) | 1 (1) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 6 (7) | 13 (21) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (25) | 18 (34) | 2 (2) | 3 (5)
Asthenia (General disorders) | 11 (18) | 18 (48) | 1 (8) | 6 (9)
Chills (General disorders) | 6 (6) | 1 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 18 (27) | 19 (31) | 3 (3) | 2 (3)
Non-cardiac chest pain (General disorders) | 4 (5) | 3 (3) | 2 (2) | 2 (3)
Oedema peripheral (General disorders) | 3 (3) | 3 (6) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 7 (8) | 3 (5) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (6) | 4 (7) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (5) | 6 (7) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 14 (23) | 17 (25) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (6) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5) | 6 (8) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 7 (9) | 2 (3) | 3 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 5 (9) | 0 (0) | 4 (6)
Tremor (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 6 (6) | 4 (7) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 3 (4) | 4 (7) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (10) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (6) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated due to business decision. No safety concerns involved in decision to terminate this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT02357147/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT02357147/SAP_001.pdf